CLINICAL TRIAL: NCT04877054
Title: Pilot Evaluation of a Telehealth Motivational Interviewing Intervention Targeting Adherence Behaviors in Youth With Sickle Cell Disease
Brief Title: Pilot Evaluation of a Motivational Interviewing Intervention Targeting Adherence Behaviors in Youth With Sickle Cell Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins All Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00285183
Record Dates: First submitted 2021-04-23; First posted 2021-05-07 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Sickle Cell Disease
Keywords: pediatric; sickle cell disease; adherence; telehealth; motivational interviewing; Hydroxyurea
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 2:1 to the intervention versus an education-only control condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Intervention sessions will occur ~once per week, with all 4 sessions being completed within 4-8 weeks. Each session will include an education and motivational interviewing (MI) component.
  Interventions: Behavioral: Adherence Treatment Program
- Education only Arm (Active Comparator): Participants in the education-only control arm will receive one education session. The education session will occur via telephone or telehealth. Education will include medication purpose and adherence strategy recommendations delivered in a single telehealth session.
  Interventions: Behavioral: Education only

INTERVENTIONS:
Behavioral: Adherence Treatment Program — 4 telehealth sessions including a combination of psycho/medical education plus a motivational interviewing component.
  Arms: Intervention Arm
Behavioral: Education only — The control group will receive an education-only session. Education will include medication purpose and adherence strategy recommendations delivered in a single telehealth session.
  Arms: Education only Arm

SUMMARY:
Sickle cell disease (SCD) is a group of inherited blood disorders affecting 100,000 individuals in the United States. SCD often leads to complications, including pain crises and organ damage. Many individuals with SCD require medications (e.g., Hydroxyurea or Endari) that research has demonstrated reduce risk of complications and improve quality of life. Despite the need for strong medication adherence, adolescents and young adults (AYAs; 13-25 years) have the lowest adherence rates compared to other age groups. Efforts to reduce AYA non-adherence risk should include youth in earlier childhood and persist throughout the AYA developmental period, with the goal of maintaining adherence throughout childhood and young adulthood. Motivational Interviewing (MI) has been effective in increasing pediatric and adult medication adherence via in-person or telehealth delivery; however, researchers have yet to empirically evaluate MI for feasibility, acceptability, and/or efficacy in improving pediatric/AYA SCD medication adherence. The proposed feasibility trial will provide preliminary feasibility data for a newly developed MI+education intervention targeting medication adherence for pediatric and adolescents and young adults (AYA) patients who have sickle cell disease. This trial will also evaluate study design feasibility to inform a future randomized controlled trial (RCT). The investigators are interested in delivering the intervention to AYA patients and to parents of younger children who have sickle cell disease because the investigators anticipate that establishing strong adherence in younger childhood could prevent future non-adherence during the AYA developmental period. Participants will include 13-22 year-old patients with sickle cell disease as well as parents of 0-22 year-old patients with sickle cell disease. The investigators will randomize ten families to a 4-session telehealth MI+education intervention and five families to a one-session education-only control condition. All participants will complete assessments at three times. Intervention participants will complete the T2 assessment at their last intervention session (week 4-8), and the T3 assessment 16-20 weeks after study enrollment. Education arm participants will complete T2 assessments 4-8 weeks after study enrollment and will complete T3 assessments 16-20 weeks after study enrollment. Primary outcomes include intervention feasibility and acceptability and study design feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Participants will include 13-22 year-old patients with sickle cell disease as well as primary caregivers of 0-22 year-old sickle cell disease patients ("parents"). The lower age limit for patients' participation in their own intervention sessions was selected based on previous studies documenting MI effectiveness with adolescents as young as 13 years of age. The upper limit was selected based on the recruitment site's (JHACH) patient population.
* Participants must be able to speak and understand spoken English because MI is language-dependent.
* The patient's SCD regimen must include at least one of the following medications: Hydroxyurea, Endari, Adakveo, or Oxbryta.
* Patients who meet inclusion criteria may participate even if their parent chooses not to do so, although 13-17 year old patients may only participate with parent consent. Likewise, parents of patients may participate even if the AYA declines their own participation, as long as the AYA assents/consents to medical chart review. Adult patients (18-22 years of age) will not require parent consent and may choose to participate with or without a parent.

Exclusion Criteria:

* Potential participants who appear to have cognitive, motor, or language delays, as observed by research personnel or documented in the medical record, will be excluded from this study if delays preclude informed consent and/or study completion. Participants may request that research personnel read all assessment, education, and intervention materials aloud in a structured interview format, in which case participants could respond to items verbally and/or by pointing to visual aids. Because of this option, participants' ability to read and write are not requirements for participation.
* Because the MI component of the intervention is language-dependent and requires significant time and training for certification in another language, non-English speaking patients will only be included in this study if the psychology postdoctoral fellow hired in this study is a native Spanish speaker and can demonstrate MI proficiency in Spanish.
* Participants who score in the clinically significant range (t-scores 2 standard deviations above the mean) on any of the PROMIS measures assessing depression and anxiety will be removed from the study and provided mental health resources.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Change in sickle cell disease medication adherence | Baseline, post intervention (weeks 4-8 after study enrollment), and 16-20 weeks after study enrollment
  This questionnaire assesses participants' adherence to their sickle cell disease medication. The questionnaire is titled Sickle Cell Antibiotic Adherence Level Evaluation (SCAALE). Question items are scored in different directions depending on whether their wording reﬂects adherence or non-adherence. For each item, participants will rate each item on a Likert scale, such that the response indicating the 'best' adherence is scored one point and the response indicating the 'worst' adherence is scored ﬁve points. Possible subscale scores range from four points (most adherent) to 20 points (least adherent),and possible total scores range from 24 (most adherent) to 120 (least adherent).
Intervention feasibility as assessed by the fidelity rating | Post intervention (weeks 4-8 after study enrollment)
  Feasibility of conducting the intervention with high clinician fidelity, as evidenced by fidelity ratings for each session (fidelity represented as a percentage based on the extent to which the clinician covered all planned information for each session). Average intervention fidelity ratings should meet or exceed 80 percent fidelity.
Intervention acceptability as assessed by the Abbreviated Acceptability Rating Profile | Post intervention (weeks 4-8 after study enrollment)
  Patient and caregiver acceptability of the newly developed intervention, as evidenced by the Abbreviated Acceptability Rating Profile. Scores range from 8-48, with higher scores indicating greater acceptability. Scores equal to or greater than 30 indicate good acceptability per published standards.

SECONDARY OUTCOMES:
Change in sickle cell disease knowledge as assessed by the Sickle-Cell Disease Knowledge Questionnaire | Baseline, post intervention (weeks 4-8 after study enrollment), and 16-20 weeks after study enrollment
  Knowledge of sickle cell disease recommendations, as evidenced by scores on the Sickle Cell Disease Knowledge Questionnaire. Scores range from 0-28, with higher scores indicate greater knowledge.
Change in healthy lifestyle self-efficacy as assessed by the Adolescent Lifestyle Profile II | Baseline, post intervention (weeks 4-8 after study enrollment), and 16-20 weeks after study enrollment
  Self-efficacy maintaining healthy lifestyle behaviors, as evidenced by scores on the Lifestyle Profile II. Total mean scores range from 1-4 with greater scores indicating greater self-efficacy.
Change in illness perception as assessed by the Brief Illness Perception Questionnaire | Baseline, post intervention (weeks 4-8 after study enrollment), and 16-20 weeks after study enrollment
  Perception of illness, as evidenced by scores on the Brief Illness Perception.Questionnaire, Total scores range from 8-10 with greater scores indicating stronger illness perception.
Change in self-esteem as assessed by the Rosenberg Self-Esteem Scale | Baseline, post intervention (weeks 4-8 after study enrollment), and 16-20 weeks after study enrollment
  Self-esteem, as evidenced by scores on the Rosenberg Self-Esteem Scale. Total scores range from 10-40, with greater scores indicating greater self-esteem.
Change in depression as assessed by the PROMIS Pediatric Depressive Symptoms-Short Form or PROMIS Adult Depressive Symptoms-Short Form | Baseline, post intervention (weeks 4-8 after study enrollment), and 16-20 weeks after study enrollment
  Depressive symptoms, as evidenced by scores on the PROMIS Pediatric Depressive Symptoms-Short Form or PROMIS Adult Depressive Symptoms-Short Form. Scores range from 1-40 with greater scores indicate greater depressive symptoms.
Change in anxiety as assessed by the PROMIS Anxiety Symptoms- Short Form or PROMIS Adult Anxiety Symptoms Short Form | Baseline, post intervention (weeks 4-8 after study enrollment), and 16-20 weeks after study enrollment
  PROMIS Pediatric Anxiety Symptoms- Short Form or PROMIS Adult Anxiety Symptoms Short Form. The adult anxiety scores range from 1-35 and the pediatric anxiety score range from 1-40 with greater scores indicate greater anxiety symptoms.
Change in health literacy as assessed by the Health Literacy Skills Instrument- Short Form for adults or the Health Literacy Assessment Scale for Adolescents (HAS-A) | Baseline, post intervention (weeks 4-8 after study enrollment), and 16-20 weeks after study enrollment
  Health literacy scores, as evidenced by scores on the Health Literacy Skills Instrument- Short Form for adults (HLSI-10) or the Health Literacy Assessment Scale for Adolescents (HAS-A). The HLSI-10 scores range from 0-10 with higher scores indicating higher levels of health literacy. The HAS-A has 3 scales. Scores on the Communication subscale range from 0-20 with higher scores representing better interpersonal communication. Scores on the Confusion subscale range from 0-16 with higher scores representing more confusion. Scores on the functional health literacy scale range from 0-20 with higher scores indicating a lower ability to read health information and understand numbers.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Faith, Principal Investigator — Johns Hopkins All Children's Hospital
Locations (1):
- Johns Hopkins All Children's Hospital, St. Petersburg, Florida, United States

IPD SHARING:
Plan to Share IPD: No